CLINICAL TRIAL: NCT03483090
Title: A Randomised, Double-blind, Placebo Controlled Study to Investigate the Effect on Knee Pain Reduction and Safety of Swisse High Strength Deep Sea Krill Oil (Superba BOOST) in Adults With Mild to Moderate Osteoarthritis of the Knee
Brief Title: Investigating the Effect of Deep Sea Krill Oil Supplementation in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swisse Wellness Pty Ltd (Industry)
Collaborators: Commonwealth Scientific and Industrial Research Organisation, Australia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUB-001
Record Dates: First submitted 2018-02-27; First posted 2018-03-30 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis, Knee
Keywords: mild; moderate; krill oil; pain; osteoarthritis; supplement
MeSH Terms: conditions — Osteoarthritis, Knee; Lymphoma, Follicular; Pain; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Treatment arm and Placebo arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): 4000mg Swisse High Strength Deep Sea Krill Oil (Superba BOOST) (4 capsules containing 1000mg each)
  Interventions: Dietary Supplement: Swisse High Strength Deep Sea Krill Oil
- Treatment B (Placebo Comparator): 4 capsules of matching Placebo orally daily (1000mg each of mixed vegetable Oil)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Swisse High Strength Deep Sea Krill Oil — Krill oil is sourced sustainably from the Southern Ocean and is extracted from the Antarctic Krill, the most abundant marine biomass. Krill oil is a source of omega-3 fatty acids, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) for the maintenance of good health. Omega-3, EPA and DHA are also found in phospholipid form which are much easier absorbed than triglyceride form of omega-3 which is found in fish oil. Omega-3 supports cardiovascular health, brain health and eye health. Preliminary research suggests krill oil can provide temporary relief from symptoms of mild arthritis, help reduce joint inflammation and increase joint mobility.
  Other Names: Superba BOOST
  Arms: Treatment A
Other: Placebo — No therapeutic effect
  Arms: Treatment B

SUMMARY:
To evaluate the effectiveness of 4 g Swisse High Strength Deep Sea Krill Oil (Superba BOOST) daily on pain reduction in adults with mild to moderate osteoarthritis of the knee compared to placebo over a 6 month period.

This is a multicentre, randomised, double-blind, placebo-controlled parallel-arm study.

Applicants will be eligible to participate if they have mild to moderate OA of the knee. Diagnosis of OA of the knee will be made according to clinical diagnosis, using the American College of Rheumatology (ACR) Criteria for the classification of Idiopathic OA of the Knee and the Kellgren-Lawrence grading scale. In addition, eligible applicants will have been experiencing knee pain on at least 4 days per week, for at least 3 months and they will report knee pain between 4 and 8 cm (inclusive) on a visual analogue scale (VAS) for the 7 days prior to Day 1 of the trial (Baseline). Severity of OA of the knee will be assessed based on X-ray performed at the Screening Visit using the Kellgren-Lawrence (KL) radiographic criteria, and participants with severe radiographic knee OA (KL joint space narrowing (JSN) above grade 3) will be excluded.

Applicants will attend a screening visit following pre-screening assessments to assess their general health and eligibility for inclusion into the study.

On Day 1 eligible participants will be randomly allocated to receive one of two study treatments. Participants will take the assigned treatments daily for six months.

Participants will return to the clinic at 3 months and 6 months for study assessments. Participants will complete an online survey at 1, 2, 4 and 5 months to assess protocol compliance, adverse events and use of concomitant medications. Any queries from the survey will be followed up by phone call.

A final participant online survey and phone call (if needed) will be conducted 28 days after the 6 month visit for a final safety assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female aged 40 - 65 years, inclusive
2. Clinical Diagnosis of OA of the index knee according to the ACR Criteria for the classification of Idiopathic OA of the Knee
3. Kellgren-Lawrence (KL) grade 1-3 OA, evidenced by Knee X-ray performed during the screening period
4. Experiencing pain of the index knee on at least 4 days per week for the last 3 months (based on self-report)
5. Pain of the index knee between 4 and 8 cm (inclusive) as self-assessed on a visual analogue scale (VAS) over the 7 days prior to Day 1
6. Body mass index (BMI) >18.5 kg/m2 and <35 kg/m2 on Day 1
7. Willingness to abstain from use of restricted medications.
8. Habitual intake of long chain (LC) omega-3 polyunsaturated fatty acids (PUFA) (from food and supplements) <500mg/day as assessed using the Australian PUFA food frequency questionnaire (FFQ) during the screening period and willingness to maintain a low intake throughout the study. Higher intakes of LC omega-3 PUFA will require a 3 month washout period.
9. Willing to provide written Informed Consent.

Exclusion Criteria:

1. Severe radiographic knee OA in any knee defined as Kellgren-Lawrence (KL) score >3 based on X-ray (weight bearing) performed during the screening period.
2. Ipsilateral hip OA such that it would compromise assessment of knee pain.
3. Fibromyalgia, chronic pain syndrome or other concurrent medical or arthritic conditions which could interfere with the evaluation of the index knee.
4. History of Reiter's syndrome, rheumatoid arthritis (RA), psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis or amyloidosis or any other forms of inflammatory arthritis (e.g. gout, pseudogout). Gout is excluded unless the participant is on preventative treatment and has not had an attack in the last 12 months.
5. History or clinical signs and symptoms of infection in the index joint in the last 5 years.
6. Knee pain that is not clinically attributable to OA of the knee (e.g., radicular low back pain and hip pain that is referred to the knee that could cause misclassification).
7. Pain in any other area of the lower extremities or back that is equal to or greater than the index knee pain (based on self-report).
8. Arthroscopy or open knee surgery in the index knee in the previous 12 months or planned for the duration of the study period.
9. Intraarticular (IA) or Intramuscular (IM) corticosteroid (investigational or marketed) in any joint within 3 months of Screening or Oral corticosteroids (investigational or marketed) within 1 month of Screening.
10. IA hyaluronic acid (investigational or marketed) in the index knee within 6 months of Screening
11. Any other IA intervention or therapy within 3 months of Screening .
12. Regular use of opioids/opiates within 4 weeks of Day 1 equivalent to >30mg codeine per day, for 5 days or more, unless participant agrees to a washout period of at least 4 weeks prior to Day 1.
13. High dose NSAIDs within the last month, defined as at the maximum dose recommended for the symptomatic treatment of arthritis pain (e.g., diclofenac ≥150 mg/day, aceclofenac ≥100 mg/day, meloxicam ≥15 mg/day, naproxen ≥1,000 mg/day, piroxicam ≥20 mg/day, and ibuprofen >2,400 mg/day), unless participant agrees to a washout period of at least 4 weeks prior to Day 1.
14. Bleeding disorders, currently taking anticoagulants or has received anticoagulants within 28 days of Day 1, with the exception of low dose aspirin up to150mg daily.
15. Regular use of and not prepared to abstain from glucosamine, fish oil, curcumin and other complementary medicines/supplements, that may affect the study results. A washout period of minimum of 4 weeks will apply prior to Day 1, except in the case of fish oil, where 3 month washout will apply.
16. Positive urine dipstick pregnancy test at screening or Day 1, currently pregnant and/or breastfeeding.
17. Women of child bearing potential (WOCBP) who:

    1. Are not currently using effective methods of contraception and
    2. have not been using effective methods of contraception for 14 days prior to Day 1 and
    3. are not willing to use effective methods of contraception throughout the study
18. History of or known presence of alcohol abuse or illicit drug use, any surgical history, clinically significant conditions (i.e renal or urological disease, cardiac disease, liver disease, gastrointestinal disease or any other significant disease) or organ dysfunction that in the opinion of the investigator may affect the participant's ability to participate in the study or the study results.
19. Currently hospitalised or any planned hospitalisations during the study or up to 1 month following the last dose of study product that may affect the participants ability to comply with the study in the opinion of the medical investigator.
20. Received an investigational drug within 3 months of Day 1 that in the opinion of the investigator may affect the applicant's ability to participate in the study or the study results.
21. Known or suspected allergies to the investigational products
22. History of an adverse reaction or known hypersensitivity to seafood or shellfish.
23. Hypertension (blood pressure ≥140/90 mmHg at screening. (Participants with an elevated BP at screening may be included if they are able to provide a treating doctor letter stating either that they do not have hypertension or that their hypertension has been well controlled for at least 4 weeks).

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome is the change in The Western Ontario and McMaster Universities Arthritis Index (WOMAC), Pain subscale (Numeric Rating Scale) | from Baseline to 6 months
  WOMAC scale is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items); Stiffness (2 items); Physical Function (17 items):
  Questionnaire scores on a scale of 0-4, None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The primary outcome related to the Pain subscale and will therefore be scored between 0 and 20.

SECONDARY OUTCOMES:
WOMAC B (stiffness subscale) change from Baseline | from Baseline to 6 months
  WOMAC scale is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items); Stiffness (2 items); Physical Function (17 items):
  Questionnaire scores on a scale of 0-4, None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  This outcome is measured on the stiffness subscale and will be therefore scored from 0 to 8.
WOMAC C (function subscale) change from Baseline | from Baseline to 6 months
  WOMAC scale is widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  Pain (5 items); Stiffness (2 items); Physical Function (17 items):
  Questionnaire scores on a scale of 0-4, None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  This outcome is measured on the physical function subscale and will therefore be scored from 0 to 68.
Serum lipid concentrations (total cholesterol, HDL-C, LDL-C, triglycerides) changes from baseline (efficacy) | from Baseline to 6 months
  Venous blood will be taken at baseline, 3 months and 6 months to measure serum cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol and triglycerides. Serum lipid variables will be measured on a Beckman AU480 clinical analyser (Beckman Coulter Inc, Brea, CA, USA) usingcommercial enzymatic test kits for Total cholesterol, triglycerides and HDL-C. LDL-C will be calculated using the Friedewald equation.
Change in inflammatory markers (IL-6, TNF-α, hsCRP) from Baseline | from Baseline to 6 months
  Venous blood will be taken at baseline, 3 months and 6 months to measure interleukin-6, tumour necrosis factor alpha and high sensitivity C-reactive protein. Serum hsCRP will be analysed using a clinical analyser and commercial assays kits (Beckman Coulter, Inc., CA, USA). Serum IL-6 and TNF-α will be analysed using the Luminex 100/200 system with xPONENT software (Luminex, Texas, USA) commercial assay kits.
Omega 3 index changes from Baseline | from Baseline to 6 months
  A finger prick dried blood spot sample will be collected for Omega 3 Index analysis using the Aker Biomarine Phlebotomy kit (ARTG 277814). The dried blood spot samples will be shipped to an accredited central clinical laboratory for analysis of fatty acids in dried blood spots and calculation of the Omega-3 Index. This will be collected at baseline, 3 months and 6 months.
Incidence of SAEs and adverse events (AEs) | from Baseline to 6 months
  Participants will be questioned, in a non-leading manner, at each visit with regard to any AEs they may have experienced since their last visit. All AEs will be recorded in source documents and will be followed until either completely resolved or until the Final Safety or Early Withdrawal visit.
Clinically significant changes in haematology from baseline | from Baseline to 6 months
  The following parameters will be measured at baseline, 3 months and 6 months: Haemoglobin, red blood cell count (RBC), Red cell distribution (RDW), Packed Cell Volume (PCV), Mean Cell Volume (MCV), Mean cell hemoglobin concentration (MCHC), Platelets, White Cell Count (WCC), Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils The medical investigator will assess deviations from laboratory reference ranges for clinical significance.
Clinically significant changes in biochemistry from baseline | from Baseline to 6 months
  The following parameters will be measured at baseline, 3 months and 6 months: Sodium, Potassium, Chloride, Bicarbonate, Glucose, Urea, Creatinine, Calcium, C reactive protein (CRP), Uric acid, Phosphate, Albumin, Globulins, Protein, Total bilirubin, Gamma-glutamyl transpeptidase (GGT), Alkaline Phosphatase (ALP), Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Lactate Dehyrogenase (LD) The medical investigator will assess deviations from laboratory reference ranges for clinical significance.
Clinically significant changes in coagulation markers from baseline | from Baseline to 6 months
  The following parameters will be measured at baseline, 3 months and 6 months: Activated partial thromboplastin time (aPTT) and Prothrombin time (PT) The medical investigator will assess deviations from laboratory reference ranges for clinical significance.
Use of concomitant medications | from Baseline to 6 months
Clinically significant changes on clinical assessments compared to baseline: vital signs | from Baseline to 6 months
  Blood pressure, pulse, respiratory rate and temperature (°C) will be measured by a designee while the participant is seated. Resting blood pressure and heart rate will be measured using an automated blood pressure monitor in a seated position after a 5-minute rest. The average of three measurements (separated by 2 minutes) will be recorded. Respiratory rate will be measured by counting the number of times the chest rises per minute while the participant is at rest. Body temperature will be measured using a digital tympanic thermometer.Vital signs will be performed at Screening, Baseline, 3 month and 6 month or Early Withdrawal Visit.
  The medical investigator will assess abnormalities for clinical significance.
Clinically significant changes on clinical assessments: physical examination | from baseline to 6 months
  A non-invasive physical examination will be performed by a Medical Investigator and will include the following outcomes: General appearance, Eyes, Ears, nose, mouth and throat, Cardiovascular, Respiratory, Gastrointestinal, Genitourinary•Musculoskeletal•SkinAt Day 1 (Baseline visit) these will be reviewed to establish their baseline characteristics. A symptom directed physical exam will be conducted at 6 months or Early Withdrawal Visit.
  The medical investigator will assess abnormalities for clinical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Welma Stonehouse, PhD, Principal Investigator — Commonwealth Scientific and Industrial Research Organisation, Australia
Locations (4):
- Australia (4):
  - University of the Sunshine Coast Clinical Trials Centre, Morayfield Health Hub, Morayfield, Queensland
  - University of the Sunshine Coast Clinical Trials Centre, USC Health Clinics, Sippy Downs, Queensland
  - CSIRO Nutrition and Health Research Clinic, Adelaide, South Australia
  - Emeritus Research, Camberwell, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stonehouse W, Benassi-Evans B, Bednarz J, Vincent AD, Hall S, Hill CL. Krill oil improved osteoarthritic knee pain in adults with mild to moderate knee osteoarthritis: a 6-month multicenter, randomized, double-blind, placebo-controlled trial. Am J Clin Nutr. 2022 Sep 2;116(3):672-685. doi: 10.1093/ajcn/nqac125. PMID 35880828